CLINICAL TRIAL: NCT06202976
Title: Mapping Epileptic Networks Using Multimodal Imaging
Acronym: CREIM
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IM-RCM-2017-02
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Epilepsy in Children
Keywords: Focal Epilepsy; Lesional Epilepsy; Nonlesional Epilepsy
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients
  Interventions: Other: Secondary data collection

INTERVENTIONS:
Other: Secondary data collection — clinical data

SUMMARY:
Currently, mapping the epileptogenic zone is based on a comprehensive preoperative assessment involving clinical, imaging and electrophysiological examinations.

To reduce the need for invasive stereoelectroencephalography (SEEG) explorations, electrophysiological and imaging methods have been developed, such as resting-state functional MRI (fMRI) coupled with electroencephalogram and arterial spin-labeling perfusion MRI (ASL-MRI).

It has been published that these new methods enable precise delineation of the epileptogenic zone and better preparation for surgery.

The aim is to determine whether, in children with focal lesional epilepsy, the combination of ASL-MRI-EEG and resting-state fMRI-EEG enables precise identification of the epileptogenic zone to be defined by SEEG, the current reference examination.

ELIGIBILITY:
Inclusion Criteria:

* Be under 18 years of age on the day of inclusion.
* Present with one of the following forms of epilepsy:

  * refractory focal lesional epilepsy
  * rare non-lesional epilepsy
* Present abnormalities (spikes) on the intercritical EEG
* Have been selected by the "Epilepsy" multidisciplinary staff.
* In the case of refractory lesional epilepsy, be required to perform an EEG-video recording using intracranial electrodes (SEEG) as part of the pre-surgical workup.
* Be affiliated to a health insurance scheme.

Exclusion Criteria:

* Requiring general anesthesia for MRI
* Require sedation specifically for research
* Have generalized epilepsy
* Be deprived of liberty or under guardianship.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with refractory focal epilepsy, possibly due to lesions
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2033-09-13 (Estimated); Study Completion 2033-09-13 (Estimated)

PRIMARY OUTCOMES:
Determine whether, in children with lesional focal epilepsy, the combination of ASL-MRI-EEG and resting-state fMRI-EEG can accurately identify the epileptogenic zone to be defined by SEEG, today's gold standard. | 15 years

SECONDARY OUTCOMES:
Study the pathophysiology of resistant lesional epilepsies | 15 years
  Measurements of perfusion in ASL-MRI (inter and/or percritical) and the BOLD effect in resting-state fMRI
Correlate cortical perfusion change on SL-ASMRI and BOLD signal abnormalities on resting-state fMRI | 15 years
Compare cortical perfusion abnormalities and resting-state fMRI based on EEG data in MRI. | 15 years
Correlate BOLD-MRI perfusion abnormalities with anatomical (DTI (tractography)) and functional (resting-state fMRI) brain connectivity abnormalities. | 15 years
Compare ASL-MRI and resting-state fMRI data coupled with EEG to the results of deep electrodes (intracranial EEG - SEEG), which are today's gold standard. | 15 years
Evaluate whether these data will eventually make it possible to reduce the frequency of intracranial EEG explorations (stereo EEG, subdural grids), with a view to replacing invasive deep electrodes in the future with multimodal MRI coupled to EEG in MRI. | 15 years
Improving understanding of the pathophysiology of rare non-lesional epilepsies | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Necker - Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No